CLINICAL TRIAL: NCT05335525
Title: Post-market Clinical Investigation of the Angio-Seal™ VIP VCD: A Prospective, Multi-center Observational Study (ANGIO-SEAL CLOSE)
Brief Title: Post-market Clinical Investigation of the Angio-Seal™ VIP VCD (ANGIO-SEAL CLOSE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Terumo Europe N.V. (Industry)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T139E4
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Vascular Closure; Endovascular Procedure; Hemostasis; Peripheral Vascular Disease; Femoral Artery
Keywords: Peripheral Intervention; CFA arteriotomy closure; Common Femoral Artery Access Site; Vascular Closude Device (VCD)
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Closure of the femoral arterial puncture site — Patient will undergo a diagnostic or interventional endovascular procedure, compatible with the use of Angio-Seal™ VIP VCD.

SUMMARY:
The present post-market surveillance study aims to evaluate the safety and effectiveness of the Angio-SealTM VIP VCD in patients undergoing endovascular procedures via femoral access in real-world setting.

DETAILED DESCRIPTION:
The proposed Post-Market Clinical Follow-up study is a prospective, multi-Center, observational study, aiming to further demonstrate the safety and effectiveness of the Angio-SealTM VIP VCD in achieving hemostasis of femoral artery access site in real-world subjects undergoing percutaneous endovascular procedures. 230 patients will be enrolled at up to 6 sites in Europe. Follow-ups are scheduled at 30 days (+7 days) by hospital visit or telephone call.

The sponsor shall provide training and the necessary guidelines to assist each investigation site on the data collection in the eCRF. Each site is responsible to report the available data requested by the CIP. In order to ensure data quality, validation & consistency, edit checks will be designed during database development. Data Management team and the study monitors will be responsible to review the data and raise queries in the eCRF. Data cleaning will be done in regular intervals specified in DMP. The final clean standardised datasets will be available prior to database lock for data analysis. An audit trail logging all data entered and edited is available within the EDC system. All source documents are maintained in the hospital files ready for inspection by the Sponsor and regulatory authorities upon request. The Sponsor will inform the investigator of the time period for retaining these records as per applicable regulatory requirements.

The study will be monitored at all stages of its development by study monitors appointed by the sponsor. Study monitors are designated as Sponsor representatives and are assigned to oversee the conduct and progress of the study at each site in accordance with the Monitoring Plan established for this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject is willing and able to complete the follow-up requirements
3. Subject has the mental capacity (i.e., does not require the use of a Legally Authorized Representative) to sign the study Informed Consent Form (ICF)
4. Patient undergoing diagnostic or interventional endovascular procedure compatible with the use of Angio-SealTM VIP VCD
5. Puncture site located at the femoral artery (i.e., between the inguinal ligament and the bifurcation of the superficial femoral and profunda femoris arteries)
6. Angio-SealTM VIP VCD deployed as per instruction for use by a trained operator

Exclusion Criteria:

* Use of the Angio-SealTM VIP VCD on puncture sites other than the femoral artery

  1. Repuncture of the femoral artery within 90 days at the same access site
  2. Lumen diameter of femoral artery < 4 mm
  3. Patients with clinically significant peripheral vascular disease at the puncture site (luminal narrowing of >40% within 5 mm of the puncture site)
  4. Puncture site at or distal to the bifurcation of the superficial femoral and profunda femoris artery
  5. Puncture site proximal to the inguinal ligament
  6. Procedure sheath placed through the superficial femoral artery into the profunda femoris
  7. Multiple femoral punctures
  8. Known or suspected posterior femoral wall puncture
  9. Use of > 8F primary introducer sheaths or devices for an 8Fr Angio-SealTM VIP, or use of a >6Fr primary introducer sheaths or devices for a 6Fr Angio-SealTM VIP
  10. Any condition that would make use of Angio-SealTM VIP VCD inappropriate (as per IFU and investigators' discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 230 enrolled subjects undergoing diagnostic or interventional endovascular procedures in which Angio-SealTM VIP VCD is used
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Successful puncture site haemostasis | 6 hours post-procedure
  Cessation of arterial bleeding (excluding oozing) achieved in the interventional lab in subjects not requiring adjunctive intervention at the access site, including manual compression.
Safety: freedom from major complications of the access site limb | 6 hours post-procedure
  Major complications attributable to Angio-Seal TM VIP VCD are defined as:
  * Access site-related bleeding (BARC type 2, 3 or 5, following Angio-SealTM VIP VCD deployment, as per Bleeding Academic Research Consortium (BARC) classification)
  * Femoral puncture site haematoma >6
  * Pseudoaneurysms requiring intervention
  * Femoral access site arteriovenous fistulas
  * Access site infection requiring hospitalization
  * Embolism (due to Anchor fracture)
  * Thrombosis at puncture site (due to collagen disposition into the artery)
  * Allergic Reaction to Angio-SealTM VIP components
  * Foreign body reaction
  * Inflammation and Edema

SECONDARY OUTCOMES:
Freedom from any minor complications at the target limb access site | 6 hours post-procedure
  Minor complications are defined as:
  * Femoral puncture site Hematoma <6cm
  * Access site Infection not requiring hospitalization
  * Pseudoaneurysm not requiring intervention
  * Vasovagal response
Freedom from any major and minor complications at the target limb access site | 30 days post-procedure
Time to hemostasis (TTH) | up to 1 day
  TTH is defined as time from completion of device deployment up to first observed arterial bleeding cessation (excluding oozing at access site) in subjects not requiring adjunctive intervention in the interventional lab
Time to ambulation (TTA) | up to 30 days
  TTA is defined as the time from device deployment up to the moment when the patient is able to ambulate
Quality of Life assessment (EQ-5D) | 30 days post-procedure
Angio-SealTM VCD usability | up to 1 day

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Hôpital Universitaire Henri Mondor, Créteil
  - Hôpital Européen Georges-Pompidou (HEGP), Interventional Radiology department, Paris
- Bonifatius Hospital Lingen, Clinic for Vascular Surgery, Lingen, Germany
- VieCuri Medisch Centrum, Venlo, Netherlands

IPD SHARING:
Plan to Share IPD: No